CLINICAL TRIAL: NCT01638273
Title: A Randomized, Open-label, Crossover Clinical Trial to Compare The Pharmacokinetics of A Pregabalin GLARS Tablet 150mg and Immediate Release Formulation After Multiple Dosing Under Fed Condition in Healthy Male Subjects
Brief Title: PK Study of Pregabalin GLARS Tablet 150mg and IR Formulation After Multiple Dosing Under Fed Condition in Healthy Male Subjects
Acronym: GLA5PR-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLA5PR-102
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Pregabalin, GLARS
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLA5PR GLARS tablet 150mg(mealed) (Experimental): Pregabalin 150mg
  Interventions: Drug: Pregabalin 150mg
- Lyrica Capsule 75mg(mealed) (Active Comparator): Pregabalin 75mg
  Interventions: Drug: Pregabalin 75mg

INTERVENTIONS:
Drug: Pregabalin 150mg — GLA5PR GLARS tablet 150mg/day(Pregabalin 150mg once a day, after meal) for three days
  Other Names: GLA5PR GLARS tablet 150mg
  Arms: GLA5PR GLARS tablet 150mg(mealed)
Drug: Pregabalin 75mg — Lyrica Capsule 150mg/day(Pregabalin 75mg twice a day, after meal) for three days
  Other Names: Lyrica Capsule 75mg
  Arms: Lyrica Capsule 75mg(mealed)

SUMMARY:
The purpose of this clinical trial is to compare the pharmacokinetic characteristics of GLA5PR GLARS tablet 150mg and Lyrica Capsule 75mg.

GLA5PR GLARS tablet 150mg is a New Formulation which is made by GL Pharm Tech.

GLARS(Geometrically Long Absorption Regulated System) is New Solution to Sustained Absorption by Extending the Absorption Site.

To overcome the shortcomings of the currently existing sustained release drug delivery technologies the investigators have recently developed a novel drug delivery system to enable a drug to be dissolved irrespective of the surrounding environment and further absorbed up to colon. The investigators coined this "Geometrically Long Absorption Regulated System(GLARS)".

DETAILED DESCRIPTION:
Basically, this system is a triple-layered tablet, comprised of upper and lower layers that swell and draw a sufficient amount of water, plus a highly water - soluble middle layer that rapidly draw water into the tablet core simultaneously.

The water drawn into the tablet (about 3 to 4 times the weight of the tablet itself) functions as an additional media which enables additional and later drug release out of the dosage form. This serves to overcome the shortage of surrounding media that has been reported to be one of the key reasons for mal-absorption of a drug in colon.

As the middle layer induces a rapid water draw into the tablet core, the penetrated water also diffuses to the upper and lower layers, which makes the tablet to rapidly swell and controls drug release.

At virtually the same time, the swollen upper and lower layers form to surround a lateral side of the middle layer, which can, in turn, further control drug release.

This relatively rigid swollen matrix structure makes drug release not affected by surrounding mechanical flux, which can provide relatively consistent in vivo drug release irrespective of degree of gastrointestinal motility.

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, Healthy Adult Male Subject
* ≥ 50kg(Body Weight) and Ideal Body Weight ≤ ±20%

Exclusion Criteria:

* ALT or AST > 1.25(Upper Normal Range)
* Total Bilirubin > 1.5 (Upper Normal Range)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cmax.ss | 36hrs
  Pharmacokinetic of Pregabalin
AUCtau | 36hrs
  Pharmacokinetic of Pregabalin

SECONDARY OUTCOMES:
Safety Monitoring | 25 days
  Adverse Event, Vital sign, Physical Exam, Laboratory Findings
Tmax | 36hrs
  Pharmacokinetic of Pregabalin
AUC0-∞ | 36hrs
  Pharmacokinetic of Pregabalin
CL/F | 36hrs
  Pharmacokinetic of Pregabalin
Vd/F | 36hrs
  Pharmacokinetic parameter of Pregabalin
T1/2 | 36hrs
  Pharmacokinetic parameter of Pregabalin

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Kim TE, Jeon JY, Gu N, Chang Kwon M, Kim MG. Comparative Pharmacokinetics of a Controlled-release Pregabalin Tablet (GLA5PR GLARS-NF1) and an Immediate-release Pregabalin Capsule in Healthy Male Volunteers. Clin Ther. 2018 Dec;40(12):2112-2124. doi: 10.1016/j.clinthera.2018.10.017. Epub 2018 Nov 27. PMID 30497798